CLINICAL TRIAL: NCT02578979
Title: Serial Electrocardiogram Versus Holter to Detect Atrial Fibrillation in Elderly Patients With Acute Ischemic Stroke: Study Protocol of a Randomized Controlled Trial
Brief Title: Serial ECG Versus Holter to Detect Atrial Fibrillation in Elderly Ischemic Stroke Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chang Gung Memorial Hospital (Other)
Collaborators: National Taiwan University Hospital (Other); Chiayi Christian Hospital (Other); Dalin Tzu Chi General Hospital (Other)
Responsible Party: Principal Investigator, Meng Lee, Associate Professor, Chang Gung Memorial Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: NMRPD1E0891
Record Dates: First submitted 2015-10-12; First posted 2015-10-19 (Estimated); Last update posted 2019-07-08 (Actual); Status verified 2019-07

CONDITIONS: Ischemic Stroke
Keywords: atrial fibrillation; ischemic stroke; electrocardiogram; holter
MeSH Terms: conditions — Ischemic Stroke; Atrial Fibrillation | interventions — Electrocardiography; Electrocardiography, Ambulatory

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- ECG for 5 days (Experimental): Patients will receive 12-lead electrocardiogram for 5 days during their hospitalization.
  Interventions: Device: Electrocardiogram
- 24-h Holter (Active Comparator): Patients will receive a 24-h Holter during their hospitalization.
  Interventions: Device: Holter

INTERVENTIONS:
Device: Electrocardiogram — Patients will receive electrocardiogram for detecting atrial fibrillation - a 5-day routine ECG.
  Arms: ECG for 5 days
Device: Holter — Patients will receive electrocardiogram for detecting atrial fibrillation - a 24-h Holter.
  Arms: 24-h Holter

SUMMARY:
Paroxysmal atrial fibrillation is often undetected because characteristics such as short duration, episodic, and frequently asymptomatic nature make it challenging to diagnose at the bedside, leading to suboptimal secondary prevention. It is not uncommon for paroxysmal atrial fibrillation to be undetected in a single electrocardiogram (ECG) on admission. Conventional 24-hour Holter monitoring is often used to detect paroxysmal atrial fibrillation. However, systematic review suggests Holter monitoring will identify atrial fibrillation in only an additional 4.6% of patients, no better than detection rates observed in groups lacking routine monitoring. On the other hand, for ischemic stroke patients with sinus rhythm at baseline but paroxysmal atrial fibrillation still suspected, no recommendation beyond repeated 12-lead ECGs is made in the United Kingdom guideline. Serial 12-lead ECG has been used to detect possible paroxysmal atrial fibrillation among acute ischemic stroke patients and found 15 new cases of atrial fibrillation in 133 acute ischemic stroke patients (11.3%) without atrial fibrillation at baseline. The optimal investigation strategy, including modality, duration of investigation, and patient subgroup remains undefined, not only for efficacy in the detection of atrial fibrillation, but also cost-effectiveness in healthcare systems. The objective of this project is to conduct a pragmatic multicenter randomized controlled trial for the comparison of serial 12-lead ECG once daily for 5 days and 24-hour Holter to detect paroxysmal atrial fibrillation in acute ischemic stroke patients without atrial fibrillation identified by baseline ECG or history.

DETAILED DESCRIPTION:
Investigators plan to enroll 900 participants from six hospitals in Taiwan. Patients will be eligible for enrollment if they are admitted due to acute ischemic stroke within 2 days, with 65 years of age or older, do not have known atrial fibrillation on history or baseline ECG at admission. Investigators will randomly assigned participants in a 1:1 ratio to undergo daily 12-lead ECG once daily for 5 days (intervention group) or 24-hour Holter monitoring (control group).

ELIGIBILITY:
Inclusion Criteria:

1. Cerebral ischemia defined as stroke (sudden focal neurologic deficit lasting >24 h consistent with the territory of a major cerebral artery and categorized as ischemic) and/or a corresponding lesion on brain imaging
2. Stroke symptoms within 2 days
3. Age ≥65 years

Exclusion Criteria:

1. History of atrial fibrillation or documented atrial fibrillation prior to randomization
2. Indication for oral anticoagulation at randomization
3. Absolute contraindication for oral anticoagulation at randomization
4. Intracerebral hemorrhage in medical history
5. Implanted pacemaker device or cardioverter/defibrillator
6. End stage renal disease

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 826 (Actual)
Dates: Start 2015-10-01 (Actual); Primary Completion 2018-07-31 (Actual); Study Completion 2018-10-31 (Actual)

PRIMARY OUTCOMES:
Number of atrial fibrillation detected | within 3 month of stroke onset

CONTACTS AND LOCATIONS:
Overall Officials: Meng Lee, MD, Principal Investigator — Chang Gung Memorial Hospital
Locations (6):
- Taiwan (6):
  - Chia-yi Christian Hospital, Chiayi City
  - Dalin Tzu Chi General Hospital, Dalin
  - Chang Gung Memorial Hospital, Keelung Branch, Keelung
  - Chang Gung Memorial Hospital, Chiayi Branch, Puzih
  - National Taiwan University Hospital, Taipei
  - Chang Gung Memorial Hospital, Linkuo Branch, Taoyuan District

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Huang WY, Lee M, Sung SF, Tang SC, Chang KH, Huang YS, Lee JD, Lee TH, Jeng JS, Chung CM, Wu YL, Hsieh TT, Ovbiagele B. Atrial fibrillation trial to evaluate real-world procedures for their utility in helping to lower stroke events: A randomized clinical trial. Int J Stroke. 2021 Apr;16(3):300-310. doi: 10.1177/1747493020938297. Epub 2020 Jul 8. PMID 32640882
- [Derived] Hsieh TT, Lee M, Huang WY, Tang SC, Sung SF, Chang KH, Lee JD, Lee TH, Huang YS, Jeng JS, Chung CM, Wu YL, Ovbiagele B. Atrial fibrillation trial to evaluate real-world procedures for their utility in helping to lower stroke events (AFTER-PULSE): Study protocol for a randomized controlled trial. Contemp Clin Trials Commun. 2017 Jun;6:127-130. doi: 10.1016/j.conctc.2017.04.005. Epub 2017 Apr 26. PMID 29082335